CLINICAL TRIAL: NCT06034652
Title: A Prospective Analysis of the Use of Gentrix® Surgical Matrix for Soft Tissue Reinforcement in Ventral Hernia Repair as Long Term Follow Up to T-GENVIH-002 Study
Brief Title: T-GENVIH-003 LTFU (Long Term Follow Up) Study
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: T-GENVIH-003
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Hernia; Hernia, Ventral; Pathological Conditions, Anatomical; Hernia, Abdominal
MeSH Terms: conditions — Hernia; Hernia, Ventral; Pathological Conditions, Anatomical; Hernia, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Prospective Analysis of Minimally Invasive Surgical Approach (i.e., laparoscopic or robotic): Collection of performance data for twenty-one subjects having prior minimally invasive surgical approach for ventral hernia repair (i.e., laparoscopic or robotic) from the previous T-GENVIH-002 study last data collection time-point (1-yr post-op) to present (prospective analysis), not previously reported.
  Interventions: Device: Integra® Gentrix® Surgical Matrix

INTERVENTIONS:
Device: Integra® Gentrix® Surgical Matrix — Integra® Gentrix® Surgical Matrix is intended for implantation to reinforce soft tissue where weakness exists in patients requiring gastroenterological or plastic & reconstructive surgery.

SUMMARY:
The T-GENVIH-003 study will collect additional, longer term performance data of Gentrix® Surgical Matrix used for reinforcement of ventral hernia repairs from a subset population (i.e., the twenty-one minimally invasive surgical approach cases) from the prior T-GENVIH-002 study.

DETAILED DESCRIPTION:
The purpose of this study is to collect additional safety data and demonstrate the performance of Integra Gentrix® Surgical Matrix for reinforcement of ventral hernia repairs from a sub-population of twenty-one participants from the previous T-GENVIH-002 study, specifically those with laparoscopic or robotic repair. Prospective data will be collected via a one-off study follow-up visit and assessed for later post-operative surgical site events and complications in the post-operative period from the last timepoint of data collection in T-GENVIH-002 to present.

ELIGIBILITY:
Inclusion Criteria:

* Patient was a subject in the T-GENVIH-002 study and underwent minimally invasive (i.e., laparoscopic or robotic) abdominal wall reconstruction for a primary hernia using Integra® Gentrix® Surgical Matrix.
* Subject has participated in the informed consent process and signed a study-specific informed consent document.
* Subject is fluent in US English or US Spanish language.
* Subject is willing to complete an e-consent and phone or in-office visit.

Exclusion Criteria:

* Not applicable.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects from the sub-population of minimally invasive surgical approach (e.g., laparoscopic or robotic) ventral hernia repair of the prior T-GENVIH-002 study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Young, PhD PMP, Study Director — Integra LifeSciences Corporation
Locations (1):
- Surgical Healing Arts, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects included in the study were from the sub-population of Minimally Invasive Surgical Approach (e.g., laparoscopic or robotic) of the T-GENVIH-002 study. No active recruitment was required.
Pre-assignment Details: Non-applicable.
Groups:
- Minimally Invasive Surgical Approach (i.e., Laparoscopic or Robotic) From GENVIH-002 Study.: Collection of performance data for twenty-one subjects having prior minimally invasive surgical approach for ventral hernia repair (i.e., laparoscopic or robotic) from the previous T-GENVIH-002 study last data collection time-point (1-yr post-op) to present (prospective analysis), not previously reported.
Period: Overall Study
Arm/Group | Minimally Invasive Surgical Approach (i.e., Laparoscopic or Robotic) From GENVIH-002 Study.
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Statistical Analysis will be based on data from all evaluable subjects meeting the eligibility criteria.
Groups:
- Sub-population of Minimally Invasive Surgical Approach of the T-GENVIH-002 Study.: Subjects in the study are from the sub-population of minimally invasive surgical approach (e.g., laparoscopic or robotic) of the T-GENVIH-002 study.
Arm/Group | Sub-population of Minimally Invasive Surgical Approach of the T-GENVIH-002 Study.
Number analyzed (Participants) | 8
Age, Continuous [Median (Standard Deviation); unit: Years] | 66.0 (13.47)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 8 out of a possible 21 pre-identified subjects (retrospective) met eligibility criteria.
  Participants
    Female | 2
    Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 5
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Confirmed Recurrence
Description: 1. Incidence of clinically confirmed recurrence of the primary hernia to date, including not previously reported in T-GENVIH-002 study.
Time Frame: Through study completion, an average of 4 months.
Population: Intent-to-Treat (ITT) Population: All subjects who are enrolled into the study provide informed consent waiver and receive study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Prospective Analysis of Minimally Invasive Surgical Approach (i.e., Laparoscopic or Robotic): Collection of performance data for eight subjects having prior minimally invasive surgical approach for ventral hernia repair (i.e., laparoscopic or robotic) from the previous T-GENVIH-002 study last data collection time-point (1-yr post-op) to present (prospective analysis), not previously reported.
  Integra® Gentrix® Surgical Matrix: Integra® Gentrix® Surgical Matrix is intended for implantation to reinforce soft tissue where weakness exists in patients requiring gastroenterological or plastic & reconstructive surgery.
Arm/Group | Prospective Analysis of Minimally Invasive Surgical Approach (i.e., Laparoscopic or Robotic)
Number analyzed (Participants) | 8
Participants | 2

2. Secondary Outcome: Self-Reported Recurrence
Description: Incidence of self-reported recurrence (i.e., bulge) of the primary hernia to date, including not previously reported in T-GENVIH-002 study.
Time Frame: Through study completion, an average of 4 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Analysis of Minimally Invasive Surgical Approach (i.e., Laparoscopic or Robotic)
Number analyzed (Participants) | 8
Participants | 3

3. Secondary Outcome: Number of Participants With Surgical Site Occurrences Requiring Procedural Intervention (SSOPI)
Description: Incidence of Surgical Site Occurrences requiring Procedural Intervention (SSOPI) of the primary hernia repair to date, including not previously reported in T-GENVIH-002.
Time Frame: Through study completion, an average of 4 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Analysis of Minimally Invasive Surgical Approach (i.e., Laparoscopic or Robotic)
Number analyzed (Participants) | 8
Participants | 1

4. Secondary Outcome: Number of Participants With Surgical Site Occurrences (SSOs)
Description: Incidence of Surgical Site Occurrences (SSOs) of the primary hernia repair to date (seroma, abscess, dehiscence, hematoma, wound necrosis, ileus, fistula, delayed wound healing), including not previously reported in T-GENVIH-002 study.
Time Frame: Through study completion, an average of 4 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Analysis of Minimally Invasive Surgical Approach (i.e., Laparoscopic or Robotic)
Number analyzed (Participants) | 8
Participants | 1

5. Secondary Outcome: Number of Subjects With Surgical Site Infections (SSIs)
Description: Incidence of Surgical Site Infections (SSIs) post primary hernia repair to date, including not previously reported in T-GENVIH-002 study.
Time Frame: Through study completion, an average of 4 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Analysis of Minimally Invasive Surgical Approach (i.e., Laparoscopic or Robotic)
Number analyzed (Participants) | 8
Participants | 1

6. Secondary Outcome: Number of Participants With Self-Reported Recurrence
Description: as for outcome 2
Time Frame: Through study completion, an average of 4 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Analysis of Minimally Invasive Surgical Approach (i.e., Laparoscopic or Robotic)
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: The safety objective is to capture existing Gentrix® Surgical Matrix Complication data in the longer term period post primary repair procedure -- to date (i.e., through study completion, an average of 4 months) -- not previously reported in T-GENVIH-002 study.
Description: [Adverse Event reporting aligns with clinicaltrial.gov definitions]
Arm/Group | Prospective Analysis of Minimally Invasive Surgical Approach (i.e., Laparoscopic or Robotic)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT06034652/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT06034652/SAP_001.pdf